CLINICAL TRIAL: NCT01666899
Title: Effect of Radiation on Tissue for Delayed Breast Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2012.032; HUM00059038 (Other: University of Michigan Medical School IRB)
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Skin and blood vessel procedures (Experimental): All patients will be placed into Arm 1. They will undergo punch biopsies of the breast skin at the time of mastectomy and at 2, 4, 6, 8 and 12 months after completion of radiation therapy. Three more biopsies will be taken at 3, 6, and 12 months after completion of reconstruction. Patients will also undergo skin blood flow studies with a laser imaging device prior to each biopsy procedure. Ultrasound studies of the chest vessels will be performed 4 times over the course of the study- once prior to radiation and at 2, 6 and 12 months after radiation.
  Interventions: Procedure: Skin and blood vessel procedures

INTERVENTIONS:
Procedure: Skin and blood vessel procedures — Biopsies, skin blood flow studies and ultrasound studies will be performed as described.

SUMMARY:
The purpose of this study is to investigate the effects of radiation therapy following mastectomy on skin and blood vessels and to use information gathered to determine an ideal time for breast reconstruction after radiation.

DETAILED DESCRIPTION:
In the setting of post-mastectomy radiation therapy delayed autologous reconstruction, favored by many attempts to avoid complications encountered with radiating the immediately reconstructed breast. The timing of delayed reconstruction is however not known. The goal of this proposal is to study the gross, structural and vascular changes in radiated mastectomy skin in addition to possible structural and flow changes of the underlying internal mammary vessels over time. We plan to use these objective findings as a basis for determining an ideal time frame for delayed autologous breast reconstruction.

Sequential mastectomy skin specimens will be obtained from 20 patients undergoing post-mastectomy radiation therapy over a 24 month period and these specimens will be evaluated histologically. These same patients will also undergo serial examinations and photographic documentation of gross skin changes. Skin perfusion will be assessed by laser Doppler imaging and internal mammary vessel structure, and flow characteristics will be assessed by color Doppler sonography.

Based on these studies, we will elucidate short and long term changes in radiated breast skin, showing inflammatory, structural and perfusion patterns that can be correlated with optimal conditions for reconstruction. This has the potential to dramatically change practice patterns of delayed reconstruction for many reconstructive surgeons and more importantly restore what patients loose with mastectomy in a consistent, timely fashion. There is also potential for improved outcomes of delayed breast reconstruction by decreasing the number of reconstructions performed too soon after completion of radiation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with invasive breast cancer who will require mastectomy and postmastectomy radiation therapy.
2. Patients who meet criteria 1, who plan on postmastectomy breast reconstruction

Exclusion Criteria:

1. Male patients
2. Patients under the age of 18
3. Patients of advanced age (greater than 75)
4. Patients with comorbidities that affect wound healing.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-10; Primary Completion 2015-06-15 (Actual); Study Completion 2015-06-15 (Actual)

PRIMARY OUTCOMES:
To evaluate cellular and histologic changes in mastectomy skin over time following completion of radiation therapy. | 2, 4, 6, 8, 12 months post radiation therapy; 3, 6, 12 months post reconstruction

SECONDARY OUTCOMES:
To evaluate the vascular density of the skin and perfusion changes following radiation therapy. | 2, 4, 6, 8, 12 months post radiation therapy; 3, 6, 12 months post reconstruction

OTHER OUTCOMES:
To evaluate changes in internal mammary vessel structure and flow characteristics over time following completion of radiation therapy. | 2, 4, 6, 8, 12 months post radiation therapy; 3, 6, 12 months post reconstruction

CONTACTS AND LOCATIONS:
Overall Officials: Adeyiza Momoh, MD, Principal Investigator — Univeristy of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States